CLINICAL TRIAL: NCT01608802
Title: Phase 3 Trial of Palliative Care for HIV Patients on Antiretroviral Therapy
Brief Title: Outcomes for Antiretroviral Therapy Patients Receiving Palliative Care
Acronym: TOPCare
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: University College, London (Other); University of Cape Town (Other)
Responsible Party: Principal Investigator, Dr Richard Harding, Associate Professor of Palliative Care, King's College London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 6594/3200
Record Dates: First submitted 2012-05-28; First posted 2012-05-31 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: HIV
Keywords: HIV; Antiretroviral therapy; Palliative care; Pain
MeSH Terms: conditions — Pain | interventions — Palliative Care; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care (Active Comparator): Standard care will be provided to the control group, i.e. existing HIV outpatient multiprofessional care, ART monitoring and adherence support.
  Interventions: Other: Standard care
- Palliative care (Experimental): Palliative care delivered by an existing nurse who has been provided with palliative care training, palliative care patient management planning records, and clinical supervision
  Interventions: Other: Palliative care

INTERVENTIONS:
Other: Palliative care — Regular appointments with an existing clinic nurse who has been trained in palliative care, the patient is asked about their physical, psychological, social and spiritual problems, and a care management plan devised with referral as necessary.
  Arms: Palliative care
Other: Standard care — Patients attend monthly for their ART monitoring and prescription filling, and a multiprofessional team is available as necessary.
  Arms: Standard care

SUMMARY:
Despite overwhelming need for effective HIV palliative care in sub-Saharan Africa, a systematic appraisal of the literature found almost no outcome or evaluative evidence.

Aim:

The investigators aim to evaluate the efficacy of HIV palliative care training and a simple palliative care assessment tool provided to nurses of patients on Antiretroviral Therapy (ART), and to evaluate this in terms of patient outcomes under clinical experimental conditions in 2 African countries using randomised controlled trial (RCT) designs.

Intervention being tested:

Within each well-established HIV ART clinic, patients will be randomly allocated to either continue receiving standard care (control group) or to receive standard care plus appointments with a clinic nurse trained in basic palliative care (intervention group).

Methods:

Design: Each Phase III clinical trial (i.e. one trial in each of 2 countries) will be powered and conducted in parallel to a common research design protocol, thus permitting evidence of outcomes that reflects 2 different ART providers, providing evidence of palliative care efficacy relevant to different HIV care settings.

Primary outcome: Each trial has been powered to a primary endpoint of pain control.

Secondary outcomes: The secondary outcomes are the core domains of palliative care as defined by the WHO (i.e. physical, including symptoms, psychological, social and spiritual) and measured by the APCA African POS. Further secondary outcomes measured will be: adherence to treatment; risk behaviours; health-related quality of life; psychological morbidity.

Inclusion: Patients will be screened and invited into the trial if they are on ART, score 3-5 on the 0-5 APCA African POS pain or symptom items, are 18 years or older, and can give informed consent to trial entry and data collection.

Analysis: An intention-to-treat analysis will be conducted to determine treatment response differences between the two conditions. In order to maximise the efficiency of longitudinal data, multi-level modelling will be applied as appropriate.

DETAILED DESCRIPTION:
Background / rationale Despite overwhelming need for effective HIV palliative care in sub-Saharan Africa (as evidenced by the epidemiology of primarily HIV and cancer), a systematic appraisal of the literature found almost no outcome or evaluative evidence. Further systematic reviews of palliative care and HIV palliative care effectiveness have found the evidence to have been generated mainly in high income countries, before the advent of antiretroviral therapy (ART) and the evidence from Africa to be of generally lower quality (i.e. non-trial data) with limited potential for inclusion in evidence-based health care planning and delivery. In order to influence clinical practice, policy and guidelines, it is essential to provide high quality trial evidence of the effectiveness of palliative care for people on ART. In order to achieve the goal of maximum coverage, the capacity building of existing HIV care services to provide palliative care to their patients seems the most feasible. Further, the evidence demonstrates that the pain and symptom burden of those on ART is not different to those not on ART, therefore a key role for palliative care may be in the support of those accessing treatment. Our proposed study will develop a model of care that extends palliative care delivery into existing HIV/ART delivery sites, offering a mechanism of greater coverage and feasibility than alternative approaches such as referral of all palliative care-related problems out to specialist external providers.

* Aim We aim to evaluate the efficacy of HIV palliative care training and a simple palliative care assessment tool provided to nurses of patients on ART, and to evaluate this in terms of patient outcomes under clinical experimental conditions in 2 African countries using randomised controlled trial (RCT) designs.
* Intervention being tested Within each well-established HIV ART clinic, patients will be randomly allocated to either continue receiving standard care (control group) or to receive standard care plus appointments with a clinic nurse trained in basic palliative care (intervention group). The intervention nurse will receive weekly supervision from a local palliative care service and will use a simple assessment form at each patient appointment.
* Methods Design: Each Phase III clinical trial (i.e. one trial in each of 2 countries) will be powered and conducted in parallel to a common research design protocol, thus permitting evidence of outcomes that reflects 2 different ART providers, providing evidence of palliative care efficacy relevant to different HIV care settings. Each of the 2 HIV care facilities (one in each of Kenya and South Africa) is a highly experienced HIV and ART care provider, with proven longevity. The providers of the palliative care training are longstanding experts in the delivery of both palliative care training and palliative care.

Primary outcome: Each trial has been powered to a primary endpoint of pain control.

Secondary outcomes: The secondary outcomes are the core domains of palliative care as defined by the WHO (i.e. physical, including symptoms, psychological, social and spiritual) and measured by the APCA African POS. Further secondary outcomes measured will be: adherence to treatment; risk behaviours; health-related quality of life; and an additional measure of psychological morbidity.

The primary and secondary outcomes are the same for each country's trial.

This study aims to reject the null hypothesis that receipt of palliative care in addition to standard care does not affect pain compared to those receiving standard care alone.

Inclusion: Patients will be screened and invited into the trial if they are on ART, score 3-5 on the 0-5 APCA African POS pain or symptom items, are 18 years or older, and can give informed consent to trial entry and data collection.

Analysis: An intention-to-treat analysis will be conducted to determine treatment response differences between the two conditions. In order to maximise the efficiency of longitudinal data, multi-level modelling will be applied as appropriate.

- Outputs We have selected an RCT design, with multiple country partners, in order that outputs have maximum potential influence.

The revised CONSORT trial statement for non-drug trials has been applied to ensure potential publication in the leading 400 medical journals.

In terms of a clinical and policy audience for the findings, the inclusion of 2 partner countries enables us to demonstrate the efficacy of 2 providers of ART care (as there is much heterogeneity between HIV care providers in Africa), and to maximise the ability to replicate findings, while dissemination will describe and compare the two providers of care delivered.

In addition to journal publications, we intend to present summary outputs to relevant Country Teams / policy / advocacy stakeholders, to present to international HIV / palliative care conference audiences, and to provide a podcast of findings to be freely downloaded on the web.

Co-applicants and Collaborators This application represents a highly effective and proven group who have, over the past 5 years, delivered clinical audit, POS tool development and validation, longitudinal studies, and various patient outcome studies in HIV palliative care in Africa. The University departments are those most closely aligned to the palliative care field in each country, and offer an active clinical / teaching / research interface. The collaboration has a strong track record of successfully conducting clinical and public health research and in clinical care. Each collaborating training palliative care centre is a long standing recognised provider of quality palliative care, operating in line with the WHO definition of palliative care.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (18 years or older),
* with an HIV diagnosis known to the patient,
* currently on ART for at least one month, and
* scoring 3-5 (out of a range of 0-5) on pain or symptoms,
* with sufficient capacity to consent to trial entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Self-report pain using the APCA African POS | Period of 4 months
  Our primary outcome is the pain item of the African Palliative Care Association Palliative care Outcome Scale

SECONDARY OUTCOMES:
Psychological morbidity | Period of 4 months
  Psychological Morbidity using the GHQ
Quality of Life | 4 month period
  Quality of Life using the MOS-HIV

CONTACTS AND LOCATIONS:
Overall Officials: Richard Harding, PhD, Principal Investigator — King's College London
Locations (2):
- BOMU Hospital, Mombasa, Kenya
- Ivan Toms Clinic, Cape Town, Western Cape, South Africa

REFERENCES:
- [Derived] Lowther K, Harding R, Simms V, Ahmed A, Ali Z, Gikaara N, Sherr L, Kariuki H, Higginson IJ, Selman LE. Active ingredients of a person-centred intervention for people on HIV treatment: analysis of mixed methods trial data. BMC Infect Dis. 2018 Jan 10;18(1):27. doi: 10.1186/s12879-017-2900-0. PMID 29316883
- [Derived] Lowther K, Selman L, Simms V, Gikaara N, Ahmed A, Ali Z, Kariuki H, Sherr L, Higginson IJ, Harding R. Nurse-led palliative care for HIV-positive patients taking antiretroviral therapy in Kenya: a randomised controlled trial. Lancet HIV. 2015 Aug;2(8):e328-34. doi: 10.1016/S2352-3018(15)00111-3. Epub 2015 Jun 15. PMID 26423375
- [Derived] Lowther K, Higginson IJ, Simms V, Gikaara N, Ahmed A, Ali Z, Afuande G, Kariuki H, Sherr L, Jenkins R, Selman L, Harding R. A randomised controlled trial to assess the effectiveness of a nurse-led palliative care intervention for HIV positive patients on antiretroviral therapy: recruitment, refusal, randomisation and missing data. BMC Res Notes. 2014 Sep 3;7:600. doi: 10.1186/1756-0500-7-600. PMID 25187211
- [Derived] Lowther K, Simms V, Selman L, Sherr L, Gwyther L, Kariuki H, Ahmed A, Ali Z, Jenkins R, Higginson IJ, Harding R. Treatment outcomes in palliative care: the TOPCare study. A mixed methods phase III randomised controlled trial to assess the effectiveness of a nurse-led palliative care intervention for HIV positive patients on antiretroviral therapy. BMC Infect Dis. 2012 Nov 6;12:288. doi: 10.1186/1471-2334-12-288. PMID 23130740
- See also: TOPCare South African launch — http://www.csi.kcl.ac.uk/topcare.html